CLINICAL TRIAL: NCT04271462
Title: The Influence of Two Different CO2 Absorbers on Sevoflurane Consumption During Anaesthesia
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Niek Sperna Weiland, Staff Anaesthesiologist (MD PhD), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W20_025 # 20.051
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing surgery (>120 min) with the use of sevoflurane based general anaesthesia (in 1.0 MAC concentration).
  Interventions: Other: Comparing two CO2 absorbers in the ventilator circuit

INTERVENTIONS:
Other: Comparing two CO2 absorbers in the ventilator circuit — General anaesthesia will be induced with a standardised regimen (propofol 0.8-2.5 mg·kg-1, sufentanil 0.2 - 0.5 µg·kg-1 and rocuronium 0.5 - 1 mg·kg-1). After tracheal intubation, anaesthesia will be maintained with sevoflurane targeted at 1 MAC end tidal concentration (corrected for age using the formula by Mapleson) in 40% O2. Different ventilator settings will be compared for 30 minutes (in randomised order):
  I. Sodalime, FGF 2.0 L min-1. II. Amsorb Plus®, FGF 2.0 L min-1. III. Soda lime, FGF, 0.5 L min-1. IV. Amsorb Plus®, FGF 0.5 L min-1. FGF=fresh gas flow.

SUMMARY:
Traditional sodalime CO2 absorbers are known to not only react with CO2 but also with sevoflurane. Therewith, a potentially harmful compound (compound A) is formed that can be nephrotoxic. In the United States, the sevoflurane manufacturer therefore recommends keeping the FGF (FGF) at >2.0 L min-1 if a sodalime CO2 absorbent is used. Amsorb Plus® (Datex-Ohmeda Inc., Madison, WI, USA), is a novel type of CO2 absorbent that does not react with sevoflurane. This allows the FGF to be reduced to 0.5 L min-1. This has two important advantages: (i) less fresh sevoflurane is added to the circle system, and (ii) the sevoflurane that is in the system does not react with the CO2 absorber.

Sevoflurane is a potent greenhouse gas with a 100 year CO2-equivalents of 120. Measures that can reduce the consumption of volatile anaesthetics could make a significant contribution to reducing the carbon footprint of the operative process. Additionally, Amsorb Plus® canisters seem to have a longer life span than sodalime canisters and do not need to be disposed of via toxic waste stream, but via domestic waste.

In this study, we were interested if (i) the use of Amsorb Plus leads to a reduction in sevoflurane usage and therefore contribute to a reduction in the CO2 footprint of general anaesthesia with sevoflurane, (ii) Does the use of Amsorb Plus® lead to a reduction in the amount of (toxic) waste produced by operating theatres?

Comparator: a traditional sodalime CO2 absorber (Medisorb™ Multi-Absorber Original, CareFusion, Helsinki, Finland).

ELIGIBILITY:
Inclusion criteria:

* Adult patient
* non-pregnant
* ASA-I to ASA-III
* undergoing Sevoflurane based general anaesthesia (in a therapeutic concentration of 1.0 MAC)
* Elective surgery
* Scheduled operating time >2 hours.

Exclusion Criteria:

* Unable/ unwilling to participate
* ASA-IV or higher
* Age < 18 years
* Known pregnancy
* Contra-indications for sevoflurane anaesthesia
* Emergency surgery
* Scheduled operating time <2 hours.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia with sevoflurane for > 2 hours.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Influence of CO2 filters on Sevoflurane consumption | 30 minutes per filter
  Comparing Sevoflurane consumption between Amsorb Plus and sodalime CO2 absorbers

SECONDARY OUTCOMES:
Influence of fresh gas flow on Sevoflurane consumption | 30 minutes per fresh gas flow setting
  Comparing Sevoflurane consumption between 0.5 and 2.0 liters per minute fresh gas flow

OTHER OUTCOMES:
Estimated CO2 footprint and environmental impact of general anaesthesia with two different CO2 filters | 30 minutes
  Estimate the CO2 footprint and environmental impact of general anaesthesia with sevoflurane comparing two different CO2 filters using life cycle analysis methods.
Estimated cost of general anaesthesia with two different CO2 filters | 30 minutes
  Estimate the total cost of general anaesthesia with sevoflurane comparing two different CO2 filters using life cycle analysis methods.
Estimated CO2 footprint and environmental impact of general anaesthesia with two fresh gas flow settings | 30 minutes
  Estimate the CO2 footprint of general anaesthesia with sevoflurane comparing two different fresh gas flow settings using life cycle analysis methods.
Estimated cost of general anaesthesia with two fresh gas flow settings | 30 minutes
  Estimate the total cost of general anaesthesia with sevoflurane comparing two different fresh gas flow settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No